CLINICAL TRIAL: NCT02664363
Title: EGFRvIII Chimeric Antigen Receptor (CAR) Gene-modified T Cells for Patients With Newly-Diagnosed GBM During Lymphopenia
Brief Title: EGFRvIII CAR T Cells for Newly-Diagnosed WHO Grade IV Malignant Glioma
Acronym: ExCeL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study funding ended
Sponsor: Daniel Landi (Other)
Responsible Party: Sponsor-Investigator, Daniel Landi, Assistant Professor of Pediatrics and Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00069444
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Results first posted 2020-07-24 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Glioblastoma; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Immunotherapy, Adoptive; Automobiles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EGFRvIII CAR T cells (Experimental): Dose escalation cohorts for 4 dose levels will be considered: #1: 4.5 x 10^6/kg, #2: 1.5 x 10^7/kg, #3: 4.5 x 10^7/kg, and #4: 1.5 x 10^8/kg. Starting at dose level 1, cohorts of 3-6 subjects will be accrued at each dose level.
  Interventions: Biological: EGFRvIII CAR T cells

INTERVENTIONS:
Biological: EGFRvIII CAR T cells — The name of the drug is CAR gene-modified T cells or abbreviated as EGFRvIII CARs. The class of action is a biological and the mechanism of action is cytotoxicity. The drug substance is autologous T cells transduced with a retroviral vector encoding for a chimeric antigen receptor (CAR) directed against the tumor specific antigen, EGFRvIII. EGFRvIII CARs are genetically engineered T cells that have been taken from patients with GBM ex vivo to express a CAR recognizing the GBM tumor-specific antigen EGFRvIII, which is expressed on a subset of GBMs but not in normal human tissues with the aim of mediating regression of their tumors. Patients' CARs will be radiolabeled with 111In for correlative studies in the expanded cohort.
  Other Names: EGFRvIII CARs; CAR-specific T cells; CAR T cells; CARs; 111Indium Labeled EGFRvIII CARs; 111In-Labeled EGFRvIII CARs; CAR gene-modified T cells; 111In-labeled CARs

SUMMARY:
Please note that enrollment on this study terminated early due to the end of grant funding.

Newly diagnosed WHO grade IV malignant glioma subjects who are eligible were enrolled following surgery to remove their brain tumor. They then underwent a leukapheresis to harvest cells for the generation of the study drug, Epidermal Growth Factor variant III Chimeric Antigen Receptor (EGFRvIII CAR) T cells prior to beginning standard of care (SOC) radiation therapy (RT) with temozolomide (TMZ). Once SOC RT with TMZ was completed, subjects returned for the post-RT brain imaging assessment, and, if stable, started post-RT TMZ cycles. Patients received up to 3 cycles of dose-intensified TMZ prior to receiving the EGFRvIII CAR T cells, which was infused in dose escalation cohorts. Following a one-month delay between cycles, the subject resumed post-RT cycles of TMZ and were monitored with blood work and brain imaging as per SOC.

An expanded cohort of 12 subjects was originally planned for once the maximally tolerated dose (MTD) was reached in the dose escalation cohorts, in order to obtain a more precise estimate of the probability of unacceptable toxicity and to track the EGFRvIII CAR T cells using 111 Indium (111In) labeling. Computed Tomography (CT) was planned on days 1, 2, and 3 post-infusion to determine intracerebral (IC) localization.

DETAILED DESCRIPTION:
Please note that enrollment on this study terminated early due to the end of grant funding.

Following consent, subjects were enrolled onto dose-escalation cohorts. Patients will underwent leukapheresis to harvest Peripheral Blood Mononuclear Cells (PBMCs) for the generation of EGFRvIII CAR T cells prior to beginning RT and concurrent TMZ. T cells were isolated from the patient's PBMCs and transduced to express the CAR. Briefly, PBMCs were stimulated with Muromonab-cluster of differentiation 3 (CD3) (OKT3), an anti-CD3 monoclonal antibody (mAb), and transduced on RetroNectin® coated plates. Transduced cells were expanded in interleukin-2 (IL-2) for 14 days.

Patients then completed standard of care RT and concurrent TMZ. Patients who remained eligible after standard of care radiation and TMZ received up to 3 cycles of TMZ at 50-100 mg/m^2/day for 21 days of 28 day cycles, which is the standard dose-intensified (DI) TMZ regimen. If the CAR-specific T cells did not meet release criteria, the patient was withdrawn before CAR treatment and replaced.

At least 48 hours after the last dose of DI TMZ, the total dose of EGFRvIII CAR T cells were delivered intravenously. If sufficient CAR-specific T cells could not be generated to meet the targeted assigned dose within the dose-escalation portion of the study, the patient was have been treated at a lower pre-defined dose level using available CAR-specific T cells and replaced in the assigned higher dose. The administered dose would have been the highest defined dose level for which there are sufficient CAR-specific T cells available. Within the expanded cohort, if sufficient CAR-specific T cells could not be generated to meet the MTD dose, all available T cells would be administered.

Following the infusion of EGFRvIII CARs, blood samples for immune monitoring were drawn 1, 5, and 10 days after the infusion, then 1, 3, and 6 months, then yearly until progression (or death or lost to contact). The return visits for immune monitoring at 3 months, 6 months, and yearly coincided with SOC clinic visits. Blood was also taken for Replication Competent Retrovirus (RCR) Polymerase Chain Reaction (PCR) per the Food and Drug Administration (FDA) at 3, 6, and 12 months during SOC clinic visits. Lastly, blood for evaluation of cytokine release syndrome (CRS) was drawn prior to cell infusion, 1 and 4 hours after infusion, and on days 1, 2, 5, 10, and at one month. Measurements for CRS included IL-2, IL-6, Tumor Necrosis Factor alpha (TNFα), interferon (IFN) gamma, Granulocyte-macrophage colony-stimulating factor (GM-CSF), and C-reactive protein (CRP).

Patients returned to clinic one month following the EGFRvIII CAR T cell infusion to be evaluated for cycles of SOC 5-day TMZ at 150-200 mg/m^2/day for the first 5-day cycle, followed by 200 mg/m^2/day for 5-days every 28 days per the treating oncologist. This resulted in a >30 day delay between the last cycle of DI TMZ and the first cycle of 5-day TMZ.

Tumor progression was documented histologically, unless there were clinical contraindications, to exclude inflammatory responses presenting as radiographic or clinical changes, which could indicate a potentially toxic or therapeutic responses and not tumor progression. If tissue was obtained through Duke Brain Tumor Center Biorepository, it was used to confirm tumor progression histologically, and to assess immunologic cell infiltration and EGFRvIII antigen escape at the tumor site. Patients would be eligible for additional adjuvant therapy at the time of tumor progression.

A classical "3+3" study design was planned to estimate the MTD for CAR-specific T cells treatment among patients with newly-diagnosed GBM. Four dose levels were to be considered: #1: 4.5 x 10^6/kg, #2: 1.5 x 10^7/kg, #3: 4.5 x 10^7/kg, and #4: 1.5 x 10^8/kg. Starting with the lowest dose level, cohorts of 3-6 subjects would be accrued at each dose level. If a patient was lost to follow-up during the first 4 weeks after CAR treatment without experiencing a dose-limiting toxicity (DLT), then the patient was not considered evaluable for the determination of DLT and would be replaced. The MTD was considered to be the highest dose level at which ≤1 of 6 patients experienced DLT during the 4-week observation period after CAR treatment. Only 3-patient cohort was enrolled at the the first dose level due to grant funding ending.

An expanded cohort of 12 patients was planned at the MTD of EGFRvIII CAR T cells, in order to obtain a more precise estimate of the probability of unacceptable toxicity. This cohort would have the cells radiolabeled with 111In to track their distribution. Briefly, CARs would have been counted and re-suspended in phosphate buffered saline (PBS). 4-6x10^8 cells would be labeled with a total of 500 microCi of 111In. The cells would be washed and mixed with cold CARs to achieve the desired cell dose. The labeled CARs would be infused into the patient through an intravenous catheter within the Ambulatory Bone Marrow Transplant (BMT) Unit. Distribution of 111In-labeled EGFRvIII CARs would be evaluated at 1, 2, and 3 days post-infusion using scintigraphy. There was no enrollment on the expanded cohort due to grant funding ending.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years of age
2. Histopathologically proven newly-diagnosed, supratentorial glioblastoma or gliosarcoma (World Health Organization [WHO] Grade IV)
3. Karnofsky Performance Status (KPS) score ≥ 70
4. The presence of the target antigen, EGFRvIII, must be identified on tumor tissue by immunohistochemistry (IHC) or Polymerase Chain Reaction (PCR).
5. Hematology:

   * Absolute Neutrophil Count (ANC) ≥ 1000/mm^3 without the support of filgrastim
   * Platelet count ≥ 100,000/mm^3
   * Hemoglobin ≥ 8.0 g/dl (eligibility level for hemoglobin may be reached with transfusion)
6. Chemistry:

   * Alanine Amino Transferase (ALT)/Aspartate Amino Transferase (AST) ≤ 2.5 times the upper limit of normal
   * Creatinine ≤ 1.6 mg/dl
   * Total bilirubin ≤ 1.5 mg/dl

Exclusion Criteria:

1. Patients who are pregnant, breast-feeding, or unwilling to practice an effective method of birth control
2. Patients with known potentially anaphylactic allergic reactions to Gadolinium-Diethylene Triamine Pentaacetic Acid (gd-DTPA)
3. Patients who cannot undergo Magnetic Resonance Imaging (MRI) or Single Photon Emission-Computed Tomography (SPECT) due to obesity or to having certain metal in their bodies (specifically pacemakers, infusion pumps, metal aneurysm clips, metal prostheses, joints, rods, or plates)
4. Patients with evidence of tumor in the brainstem, cerebellum, or spinal cord, or with evidence of leptomeningeal disease
5. Active infection requiring treatment or an unexplained febrile (> 101.5 F) illness
6. Known autoimmune disease, immunosuppressive disease or human immunodeficiency virus (HIV) infection (i.e., known HIV or Hepatitis C)
7. Patients with unstable or severe intercurrent medical conditions such as severe heart or lung disease
8. Patients with previous history of radiosurgery, brachytherapy, gliadel implantation, or radiolabeled monoclonal antibodies
9. Prior antitumor therapy for glioma (other than steroids)
10. Allergic to TMZ

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2019-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ashley, MBBS, FRACP, PhD, Principal Investigator — Duke University Hospital; Daniel Landi, MD, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suryadevara CM, Desai R, Abel ML, Riccione KA, Batich KA, Shen SH, Chongsathidkiet P, Gedeon PC, Elsamadicy AA, Snyder DJ, Herndon JE 2nd, Healy P, Archer GE, Choi BD, Fecci PE, Sampson JH, Sanchez-Perez L. Temozolomide lymphodepletion enhances CAR abundance and correlates with antitumor efficacy against established glioblastoma. Oncoimmunology. 2018 Feb 21;7(6):e1434464. doi: 10.1080/2162402X.2018.1434464. eCollection 2018. PMID 29872570

RESULTS

PARTICIPANT FLOW:
Groups:
- EGFRvIII CAR T Cells: 4.5 x 10^6 EGFRvIII CAR T Cells/kg - Autologous T cells transduced with a retroviral vector encoding for a chimeric antigen receptor (CAR) directed against the tumor specific antigen, EGFRvIII
Period: Overall Study
Arm/Group | EGFRvIII CAR T Cells
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- EGFRvIII CAR T Cells: 4.5 x 10^6 EGFRvIII CAR T Cells/kg: Autologous T cells transduced with a retroviral vector encoding for a chimeric antigen receptor (CAR) directed against the tumor specific antigen, EGFRvIII
Arm/Group | EGFRvIII CAR T Cells
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.33 (3.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximally Tolerated Dose
Description: Within this "3+3" phase I study, the primary objective is to determine the MTD of a single IV infusion of EGFRvIII CAR T cells in patients with newly-diagnosed WHO grade IV malignant glioma. Four dose levels were to be considered based on transduced cells/kg: #1: 4.5 x 10^6/kg, #2: 1.5 x 10^7/kg, #3: 4.5 x 10^7/kg, and #4: 1.5 x 10^8/kg. The MTD is the highest dose level at which ≤1 of 3-6 patients experience dose-limiting toxicity during the 4 weeks after CAR infusion.
Time Frame: 12-18 months
Population: All patients who received EGFRvIII CAR T cells
Measure: Number; unit: Cells/kg
Arm/Group | EGFRvIII CAR T Cells
Number analyzed (Participants) | 3
Cells/kg | NA — The study terminated before a MTD could be determined.

2. Secondary Outcome: Number of Patients Who Experienced a Dose-limiting Toxicity (DLT)
Description: DLT is defined as any Grade IV event of any duration that is at least (possibly, probably, or definitely) attributable to EGFRvIII CARs, or any Grade III toxicity that is at least (possibly, probably, or definitely) attributable to EGFRvIII CARs that is not reversible within 4 weeks.
Time Frame: 12-18 months
Population: All patients who received EGFRvIII CAR T cells
Measure: Count of Participants; unit: Participants
Arm/Group | EGFRvIII CAR T Cells
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | EGFRvIII CAR T Cells
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EGFRvIII CAR T Cells (N=3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EGFRvIII CAR T Cells (N=3)
Anemia (Blood and lymphatic system disorders) | 1
Eye disorders - Other, Specify: DOUBLE VISION, INTERMITTENT (Eye disorders) | 1
Vitreous hemorrhage (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Gait disturbance (General disorders) | 2
Infections and infestations - Other, Specify: FUNGUS FEET AND GROIN (Infections and infestations) | 1
Infections and infestations - Other, Specify: RING WORM (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Skin and subcutaneous tissue disorders - Other, Specify: FLUSHED/REDNESS (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT02664363/Prot_SAP_000.pdf